CLINICAL TRIAL: NCT00997217
Title: The Effect of Remote Ischemic Preconditioning on Mortality and Morbidity in Cardiac Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Remote Ischemic Preconditioning in the Cardiac Surgery
Acronym: RIPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Jeon, YunSeok, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RIPCmulticenter
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Myocardium; Injury; Cardiac Surgical Procedures
Keywords: RIPC; cardiac surgery; ischemic preconditioning; cardiac surgical procedures
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: remote ischemic preconditioning — remote ischemic preconditioning (4 x 5 min upper limb ischemia with pneumatic cuff up to 200 mmHg with an intervening 5 min reperfusion; 2 cycles; before and after the coronary anastomosis or cardiopulmonary bypass)
  Other Names: Blood pressure pneumatic cuff

SUMMARY:
Perioperative myocardial injury is a serious complication of cardiac surgery. This complication increases both mortality and morbidity of cardiac surgery. Remote ischemic preconditioning (RIPC) is the concept that brief ischemia followed by reperfusion in an organ can reduce subsequent ischemia-reperfusion injury in distant organs. Recent several clinical trials showed powerful myocardial protective effect of remote ischemic preconditioning by reducing postoperative cardiac enzymes. However, the evidence that remote ischemic preconditioning can improve the clinical outcomes such as mortality and morbidity, is still lacking. The investigators perform a multicenter randomized controlled study to evaluate that remote ischemic preconditioning can improve the outcomes of cardiac surgery.

DETAILED DESCRIPTION:
Perioperative myocardial injury is a serious complication of cardiac surgery. This complication increases both mortality and morbidity of cardiac surgery. Remote ischemic preconditioning (RIPC) is the concept that brief ischemia followed by reperfusion in an organ can reduce subsequent ischemia-reperfusion injury in distant organs. Recent several clinical trials showed powerful myocardial protective effect of remote ischemic preconditioning by reducing postoperative cardiac enzymes. However, the evidence that remote ischemic preconditioning can improve the clinical outcomes such as mortality and morbidity, is still lacking. The investigators perform a multicenter randomized controlled study to evaluate that remote ischemic preconditioning can improve the outcomes of cardiac surgery.

Purpose:

The purpose of this study is to examine if remote ischemic preconditioning can decrease the mortality and fatal postoperative complications in patients undergoing cardiac surgery. The effect will be assessed by mortality, severe morbidities and duration of hospital stay.

Methods:

Study patients will be randomized to cardiac surgery with RIPC or conventional cardiac surgery in two cardiac surgical centers (Seoul National University Hospital and Asan Medical Center). Remote ischemic preconditioning consists of four 5 min cycles of upper limb ischemia and reperfusion with pneumatic cuff up to 200 mmHg. RIPC is performed twice: before and after the coronary anastomosis in off-pump coronary bypass graft surgery; or before and after the cardiopulmonary bypass in the cardiac valve surgery.

Primary study outcome is in-hospital death within 30 postoperative days and fatal postoperative complications such as myocardial infarction, stoke, respiratory failure, renal failure, cardiogenic shock and gastrointestinal complications. Secondary outcomes include the length of intensive care unit (ICU) stay and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing cardiac surgery

Exclusion Criteria:

* emergent operation
* preoperative use of inotropics or mechanical assist device,
* left ventricular ejection fraction less than 30%,
* severe liver, renal and pulmonary disease,
* recent myocardial infarction (within 7 days),
* recent systemic infection or sepsis (within 7 days)
* peripheral vascular disease affecting upper limbs
* amputation of the upper limbs
* major combined operation such as aortic surgery or carotid endarterectomy
* descending thoracic aortic surgery
* rare surgeries; cardiac transplantation, correction of complicated congenital anomalies, pulmonary thromboembolectomy, etc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
In-hospital death | Postoperative 30 days
Myocardial infarction | Postoperative 30 days
Stroke | Postoperative 30 days
Respiratory failure | Postoperative 30 days
Renal dysfunction | Postoperative 30 days
Renal failure | Postoperative 30 days
Cardiogenic shock | Postoperative 30 days
Gastrointestinal complication | Postoperative 30 days

SECONDARY OUTCOMES:
Length of ICU stay | Postoperative 3 months
Length of postoperative hospital stay | Postoperative 3 months

CONTACTS AND LOCATIONS:
Overall Officials: YunSeok Jeon, professor, Study Director — Department of Anesthesiology and Pain Medicine, SNUH
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho YJ, Lee EH, Lee K, Kim TK, Hong DM, Chin JH, Choi DK, Bahk JH, Sim JY, Choi IC, Jeon Y. Long-term clinical outcomes of Remote Ischemic Preconditioning and Postconditioning Outcome (RISPO) trial in patients undergoing cardiac surgery. Int J Cardiol. 2017 Mar 15;231:84-89. doi: 10.1016/j.ijcard.2016.12.146. Epub 2016 Dec 23. PMID 28043669
- [Derived] Hong DM, Lee EH, Kim HJ, Min JJ, Chin JH, Choi DK, Bahk JH, Sim JY, Choi IC, Jeon Y. Does remote ischaemic preconditioning with postconditioning improve clinical outcomes of patients undergoing cardiac surgery? Remote Ischaemic Preconditioning with Postconditioning Outcome Trial. Eur Heart J. 2014 Jan;35(3):176-83. doi: 10.1093/eurheartj/eht346. Epub 2013 Sep 7. PMID 24014392